CLINICAL TRIAL: NCT06375681
Title: Examining the Effectiveness of Cognitive Training
Brief Title: Effectiveness of Cognitive Training in Older and Younger Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-1378: R01; 1R01AG076157-01 (NIH); A487400 (Other: UW Madison)
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change
Keywords: Cognitive Training; Training task; Testing context

STUDY DESIGN:
Intervention Model Description: Following Pre-testing, participants randomly assigned into the full study will be further randomly assigned to a total of 9 unique experimental conditions for the full 2x2x2+1 factorial design.
  The full description of the study's 9 arms will be registered after data collection is completed to preserve the scientific integrity of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: All researchers that have contact with participants will be unaware of the tested hypothesis of the study.
  Participants will be unaware of the experimental conditions.
  Researchers and participants will be unaware (blinded) to the game conditions assigned to the participant, except for researchers in charge of supervising the training part of the study who will be aware what training the participant is undergoing.
  More information on how this was achieved will be registered after data collection is completed to preserve the scientific integrity of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Testing Group (Active Comparator): Participants will go through 2 assessment sessions over 2-3 days (~75 minutes each), followed by 1 session of 75 minutes about 2 weeks later, 2 further sessions (~75 minutes) over 2-3 days about 2 weeks after this session, and finally another 2 sessions (~45 minutes) 3 days to 2 weeks after that session. Sessions might take place either at home or in the lab.
  Interventions: Behavioral: Visual and / or Auditory Cognitive Tasks (1)
- Long Testing Group (Active Comparator): Participants will go through 2 assessment sessions over 2-3 days (75 minutes each), followed by 10 sessions of cognitive tasks over 2 weeks, 1 session of 75 minutes about 2 weeks later, another 10 sessions of cognitive tasks over 2 weeks, then 2 sessions (~75 minutes) over 2-3 days about 2 weeks after this session, and finally another 2 sessions (~45 minutes) 3 days to 2 weeks after that session. Sessions might take place either at home or in the lab.
  Interventions: Behavioral: Visual and / or Auditory Cognitive Tasks (1); Behavioral: Visual and / or Auditory Cognitive Tasks (2)

INTERVENTIONS:
Behavioral: Visual and / or Auditory Cognitive Tasks (1) — Seven sessions (~45-75 minutes) of cognitive tasks in the lab.
  Participants asked to view visual stimuli (such as black and white lines, letters, simple shapes like triangles, circles, and squares) presented on a computer or television screen and/or listen to auditory stimuli (such as pure tones) presented via headphone or speakers and asked to make simple judgements.
Behavioral: Visual and / or Auditory Cognitive Tasks (2) — Two sets of 10 sessions (~20 minutes) of cognitive tasks either at home or in the lab.
  Participants asked to view visual stimuli (such as black and white lines, letters, simple shapes like triangles, circles, and squares) presented on a computer or television screen and/or listen to auditory stimuli (such as pure tones) presented via headphone or speakers and asked to make simple judgements.
  Arms: Long Testing Group

SUMMARY:
The proposed study will enroll 1600 participants to examine the effectiveness of cognitive training. Participants will be randomized into different experimental groups and can expect to participate for up to 15 hours of research over 4 to 8 weeks.

DETAILED DESCRIPTION:
Participants will first complete two sessions (~75 minutes each) where they are asked to view visual stimuli (such as black and white lines, letters, simple shapes like triangles, circles, and squares) presented on a computer or television screen and/or listen to auditory stimuli (such as pure tones) presented via headphone or speakers. They will be asked to make some simple judgments about the stimuli (such as indicating whether the stimulus you observed is the same or different from that on a previous trial), and indicate their judgment decision with a button press on a keyboard, a mouse click, or a movement on a touchpad. They will also be asked to complete a set of questionnaires.

After the initial sessions, participants may be asked to complete two sets of 10 sessions (~20 minutes) of cognitive tasks either at home or in the lab. Each set of sessions should be completed over a period of no more than 15 days. If asked to do these sessions, instructions will be given regarding the tasks to complete in these training sessions (which will be similar to some of the tasks you complete in the first two sessions, ~20 minutes) prior to these sessions.

After completing the first set of 10 sessions, participants will complete, either at home or in the lab, one session (~75 minutes) of tasks similar to the first sessions. Participants who were not asked to complete the 20-minute sessions will complete another session two weeks after the first two 75-minute sessions in the same location as they completed the two 75-minute sessions.

Then, participants will complete the second set of ten 20-minute sessions, or wait for about two weeks for those not asked to complete the 20-minute sessions of cognitive tasks. After this, participants will complete two other sessions (~75 minutes) in the same location as they completed the previous two 75-mintue sessions.

Finally, after a couple of weeks, participants will complete their two final testing sessions (~45 minutes each) in the same location as they completed the previous two 75-mintue sessions.

The total duration of the study will be around 8 hours if not asked to complete the twenty 20-minute sessions, or 15 hours if asked to complete these sessions. The whole experiment runs over the course of 4 to 8 weeks.

*To maintain scientific integrity, certain details of this study will not be shared until all data has been collected.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported normal or corrected-to-normal vision
* No known neurological impairments

Exclusion Criteria

* Abnormal visual acuity prohibitive of training
* History of seizures, focal brain lesion, or head injury with loss of consciousness in the past year
* Physical handicap (motor or perceptual) that would impede training procedures
* Medical illness requiring treatment during the study timeline
* Social, educational or economic hardship prohibitive to training schedule
* Concurrent enrollment in other cognitive training studies
* History of major psychiatric illness, including psychosis, bipolar disorder, alcohol or substance abuse, recent bereavement
* Score of 5 or more (i.e. presence of mild, moderate, or severe depression) on the Patient Health Screening Questionnaire (PHQ-9 Depression Screening); any participants reporting suicidal tendencies will be immediately referred to the site-specific Emergency Psychiatry Services (24-hour availability), and those with high depressive symptoms will be referred to their personal physician
* Current alcohol consumption that exceeds 14 drinks per week
* Illicit drug use
* Plans to travel out of the area for more than 1 week during the intervention period
* Residence too far from the testing site, which would prevent attending the testing sessions (> 60 miles)
* Not being proficient enough in English that would prevent following and understanding all instructions and completing all testing sessions (typically, participants would need to have learned English before age 11; there might be some exceptions that will be decided on a case-by-case basis).

Additional exclusion criteria for older adults:

* Diagnosis of dementia or other neurological disease, including mild cognitive impairment (MCI)
* Score < 26 (out of 30) on the Mini Mental State Exam (MMSE)
* Score < 18 (out of 22) on the Telephone Montreal Cognitive Assessment (T-MoCA).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in the difference between the proportion of hits minus false alarms for a given level of the N-back task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The n-Back Task is a measure of working memory. The participant is sequentially shown a series of letters and is asked to indicate whether the current letter matches the letter presented "n" items before. The n levels range between 1- and 4-back. Each level of n-back has 17-19 letters, with 5 target letters.
Change in the proportion of correctly reported sequences in the Corsi Complex task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The Corsi Complex Task is a measure of working memory. The participant is sequentially shown a series of positions from 12 possible predefined spots on the screen. Between each position, the participants is also asked to categorize a stimulus between two categories based on color and shape. The participant's task is to report the sequence of positions in order. The length of sequence can vary between 2 and 10.
Change in the proportion of correctly reported number and letter sets in the Letter-Number task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The Letter-Number Sequence Task is a measure of working memory. In each trial, the participant is presented with a sequence of alternating letters and numbers, from 2 to 10 stimuli. Participants have to report the numbers in ascending order, and the letters in alphabetical order.
Change in the difference of response time and accuracy in switch trials minus non-switch trials in the Task Switching Task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The Task Switching task is a measure of cognitive flexibility. On each trial, participants view a letter and a digit. A cue tells the participant to either categorize the letter as a consonant or vowel or else categorize the digit as even or odd. Trials can be either "non-switch trials" - in which the participant is asked to perform the same task as on the previous trial - or "switch trials" - in which the participant is asked to perform the opposite task as on the previous trial. The participant will complete 48 trials. A "switch cost" is calculated by subtracting the average response time for switch trials from the average response time for non-switch trials.
Change in the difference of response time in (i) switch trials minus non-switch trials and (ii) congruent minus incongruent trials in the Flanker Task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  In the Flanker task, the participant is asked to indicate whether the centrally presented arrow is pointing either to the left or right by pressing the left or right triangular buttons. This arrow is surrounded by 4 identical arrows, 2 to its left and 2 to its right; these are called non-target arrows. The participant is presented with two different trial types during the task, incongruent and congruent. In the congruent trials, the non-target arrows point in the same direction as the target arrow (e.g. all to the left) and in the incongruent trials they point in the opposite direction (e.g. target to the right, non-targets to the left). Switch trials are trials preceded by a trial of the opposite category (i.e. congruent preceded by incongruent or incongruent preceded by congruent).
Change in the proportion of correctly identified targets in the mixed condition of the Cancellation task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The Cancellation task is a measure of cognitive flexibility. Participants are presented with rows of 8 stimuli that can be either cats or dogs. Each cat and dog varies along its orientation, color pattern, and/or stance, giving 4 distinct cats and 4 distinct dogs. One cat and one dog are targets, and the rest are distractors. The goal of the participant is to mark as many targets as possible within each row in the allotted time (210 seconds).
Change in the proportion of correct responses on the Useful Field of View (UFOV) Task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The UFOV is a measure of visual selective attention. Participants are briefly presented with a display consisting of 24 peripheral items (3 on each of the four radial spokes and the four obliques; evenly spaced) and 1 central stimulus (a smiley with either long or short hair). One of the peripheral items is a target, while the remaining items are distractors. The participants' task is to indicate upon which of the 8 spokes the target appeared, and whether the central smiley had short or long hair. The display times vary between 16-500ms.
Change in the proportion of correct responses on the Multiple Object Tracking (MOT) Task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The MOT is a measure of visual divided attention. On each trial, participants view a series of blue and yellow smiley faces randomly moving in circular area. After a few seconds, the blue faces become yellow, indistinguishable from the distractors, while all the items keep moving on the screen. After another period of a few seconds, the items stop, and the participant is asked whether a randomly selected face was initially blue or yellow at the beginning of the trial.
Change in the response time and percentage of correct responses in the Mental Rotation Task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The mental rotation task is a measure of spatial cognition. Each trial displays two 2-D images, and the participant is asked whether the image on the right is a rotated version or a mirror-reserved and rotated version of the image on the left. The participant will complete 36 trials.
Change in the percentage of correct responses in the Paper Folding task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The Paper Folding task is a measure of mental rotation. Participants are shown 2-4 images depicting a piece of paper being folded with a hole being punched after the last fold. The participant is asked to imagine and indicate what the paper would look like unfolded. The participant will complete 10 trials.
Change in the sum of correctly solved items in Raven's Advanced Progressive Matrices task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  Raven's Advanced Progressive Matrices task is a measure of fluid intelligence. The participant is presented with a grid of elements with one of the elements missing and is asked to identify the missing element that completes the grid pattern. The participant will complete 14 trials.
Change in the sum of correctly solved items in the UC Matrix Reasoning task | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  The UC Matrix Reasoning task is a measure of fluid intelligence. The participant is presented with a grid of elements with one of the elements missing and is asked to identify the missing element that completes the grid pattern. The participant will complete 16 trials.
Change in the percentage of accuracy in the Shipley Institute of Living Scale | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  Participants will complete Part I of the Shipley Institute of Living Scale, which is a measure of vocabulary. Participants are asked to select the appropriate synonym for a target word among several alternatives for 15 words.
Change in the percentage of accuracy in the Mill-Hill Vocabulary Scale | Pre-test (baseline), post-test1 up to 30 days, (unmasked) post-test2 up to 60 days
  In this vocabulary task, participants are asked to select the appropriate synonym for a target word among several alternatives for 25 words.

SECONDARY OUTCOMES:
Big-5-Inventory 10-item version (BFI-10) Score | Pre-Test
  Individual differences in personality moderating the potential link between expectations and performance on the battery of cognitive tasks. BFI-10 measures the individuals' personality traits: conscientiousness, agreeableness, neuroticism, openness to experience, and extraversion. The total possible range of scores is from 1-5 for each personality traits, where higher scores indicate higher expression of this personality trait.
Behavioral Inhibition/Activation System (BIS/BAS) Score | Pre-Test
  Individual differences in reward sensitiveness moderating the potential link between expectations and performance on the battery of cognitive tasks. BIS/BAS measures the sensitivity to reward through four components, one inhibition component (punishment sensitivity) and three activation components (fun seeking, reward responsiveness, and drive). The total possible range of scores is from 1-4, where higher scores indicate higher expression of each dimension of the questionnaire.
Grit and Conscientiousness Score | Pre-Test
  Individual differences in grit and conscientiousness moderating the potential link between expectations and performance on the battery of cognitive tasks. Grit and Consciousness measures the tendency to sustain effort toward long-term goals. The total possible range of scores is from 1-5, where higher scores indicate higher levels of grit and conscientiousness.
Meta-Cognition Score | Pre-Test
  Individual differences in meta-cognitive skills moderating the potential link between expectations and performance on the battery of cognitive tasks. Meta-Cognition measures the ability to understand one's own abilities, strengths, and weaknesses. The total possible range of scores is from 1-5, where higher scores indicate higher meta-cognitive skills.
Theories of Intelligence - Mindset (Fixed vs Growth) Score | Pre-Test
  Individual differences in mindset moderating the potential link between expectations and performance on the battery of cognitive tasks. Theories of Intelligence - Mindset (Fixed vs Growth) measures the extent to which the participants believe that intelligence is fixed or malleable. The total possible range of scores is from 1-4, where higher scores indicate a stronger endorsement of the growth mindset than a fixed mindset, and lower scores a stronger endorsement of the fixed mindset than a growth mindset.
Schutte self-report emotional intelligence test (SSEIT) Score | Pre-Test
  Individual differences in emotional intelligence moderating the potential link between expectations and performance on the battery of cognitive tasks. SSEIT measures the ability to know and understand both one's own emotions and the emotions of others. The total possible range of scores is from 1-5, where higher scores indicate higher emotional intelligence.
Work and Family Orientation (WOFO) Score | Pre-Test
  Individual differences in achievement motivation moderating the potential link between expectations and performance on the battery of cognitive tasks. WOFO is a measure the achievement motivation of participants on three separate scales: one for work (positive attitudes toward hard work), one for general mastery (preference for difficult, challenging tasks), and one for competitiveness. The total possible range of scores is from 1-5 for each dimension of the questionnaire, where higher scores indicate more positive attitudes toward hard work, higher preference for difficult, challenging tasks, and higher competitiveness respectively.
Brief Pittsburgh Sleep Quality Index (B-PSQI) Score | Pre-Test
  Individual differences in sleep quality moderating the potential link between expectations and performance on the battery of cognitive tasks. B-PSQI is a measure the overall sleep quality of participants. The total possible range of scores is from 0-15, where higher scores indicate worse sleep quality.
Participant Experience Measure 1 | End of Post-Test (up to 60 days)
  Measure will be scored from 0-5 and will be revealed when participant data collection is completed.
Participant Experience Measure 2 | End of Post-Test (up to 60 days)
  Measure will be scored from 0-5 and will be revealed when participant data collection is completed.
Participant Experience Measure 3 | End of Post-Test (up to 60 days)
  Measure will be scored from 0-5 and will be revealed when participant data collection is completed.
Participant Experience Measure 4 | Beginning of Post-Test (up to 60 days)
  Measure will be scored from 0-5 and will be revealed when participant data collection is completed.
Participant Experience Measure 5 | Beginning of Post-Test (up to 60 days)
  Measure will be scored from 0-7 and will be revealed when participant data collection is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R. Seitz, PhD, Principal Investigator — University of California, Riverside; Susanne M. Jaeggi, PhD, Principal Investigator — Northeastern University
Locations (3):
- United States (3):
  - University of California, Riverside, Riverside, California
  - Northeastern University, Boston, Massachusetts
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (anonymized).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria.

DOCUMENTS (1):
  • Informed Consent Form (2025-11-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT06375681/ICF_000.pdf